CLINICAL TRIAL: NCT05108090
Title: Sentinel Lymph Node Biopsy for Cutaneous Squamous Cell Carcinoma of the Head and Neck
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jessica Yesensky, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CTO-OTHN-IUSCC-0741
Record Dates: First submitted 2021-10-10; First posted 2021-11-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma; Nonmelanoma Skin Cancer; Cutaneous Squamous Cell Carcinoma
Keywords: sentinel lymph node biopsy
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Procedure/Surgery (Other): Mohs micrographic surgery followed by sentinel lymph node biopsy
  Interventions: Procedure: sentinel lymph node biopsy (SLNB)

INTERVENTIONS:
Procedure: sentinel lymph node biopsy (SLNB) — Preoperative Lymphoscintigraphy: A standard injection of 2 mCi of 99m-Technetium sulfur colloid. Sequential immediate and delayed images will be obtained using SPECT/CT using a gamma probe. Ten-second counts will be done in areas of high activity to identify location of sentinel lymph node (SLN). After removal of the lymph node, a 10-second count will be done of the lymph node ex-vivo followed by 10-second count of the lymph node resection bed to ensure removal of SLN (less than 10% activity of LN).
  Surgical resection: Mohs micrographic surgery followed by SLNB. Intraoperative margins around the tumor will be confirmed through frozen section analysis. Patients with planned free flap reconstruction, will undergo SLNB with intraoperative, frozen section analysis. If lymph node is positive, immediate completion neck dissection will occur.

SUMMARY:
The purpose of this study is to research if a type of biopsy known as sentinel lymph node biopsy (SLNB) can help in determining the rate of tumor deposits that are hard to detect and identify in node-negative cutaneous squamous cell carcinoma of the head or neck.

DETAILED DESCRIPTION:
Nonmelanoma skin cancer is the most commonly diagnosed malignancy in the United States, with cutaneous squamous cell carcinoma (cSCC) representing about 20% of those cases. It is estimated that there are 700,000 patients diagnosed each year in the United States and the incidence has been increasing worldwide. Most tumors are found within the sun-exposed areas of the head and neck. The vast majority require only local treatment, however there is a subset of patients who present with regionally metastatic disease. Retrospective reviews have determined factors associated with recurrence, metastasis, and disease-specific death include tumor size ≥ 2 cm, location on lip and ear, perineural and lymphovascular invasion, poorly differentiated histology, tumor extension beyond fat and immunosuppressed patients.

There have been multiple proposed staging schemes, including the American Joint Committee on Cancer (AJCC) and recently the Brigham and Women's Hospital (BWH) tumor staging. AJCC staging utilizes the size for early stage tumors, T1 < 2 cm and T2 ≥ 2 cm and less than 4 cm. Advanced tumors, T3 and T4 are stratified by aggressive features, including invasion beyond fat, perineural invasion (PNI), or bone/skull base erosion. BWH aimed to better stratify tumors by the number of aggressive features, T1 tumors with 0 features, T2a tumors with 1 feature, T2b with 2-3 features, and T3 with 4 or more features. High-risk features include tumor diameter ≥ 2 cm, poorly differentiated histology, PNI, tumor invasion beyond fat, or bone erosion. In a recent study, and found BWH provided superior prognostication for patients with localized cSCC as compared to AJCC7. However, BWH does not address regional or distant metastasis and therefore current treatment guidelines are based on BWH staging scheme. AAJCC systemCurrently, there is a general paucity of prospective data that can provide a consensus on risk-stratification of cutaneous squamous cell carcinomas and subsequent treatment algorithm. A consensus on risk-stratification for high-risk cSCC is lacking; consequently, treatment algorithm for primary tumors and nodal disease is not clear.

There is a subset of tumors with increased risk of local recurrence, nodal and distant metastasis which has yet to be elucidated. Data has shown metastasis to regional lymph nodes is the strongest predictor of recurrence and survival, and risk of nodal metastasis is noted to be 6% for all-comers and upwards of 20% for high-risk tumors. Therefore, detecting subclinical metastatic disease is extremely important for staging aggressive skin cancers and optimizing treatment.Imaging, including CT, MRI and PET, are considered for high-risk tumor. Data has demonstrated a higher risk of developing local recurrence, nodal metastasis and death from disease in patients that did not receive pre-treatment imaging as compared those who underwent imaging.

Guidelines recommend surgical excision of the primary tumor as first line treatment for cutaneous squamous cell carcinoma. Both Moh's micrographic surgery (MMS) and standard excision are both considered feasible surgical options. Available literature on management of lymph node metastasis largely limited to retrospective reviews and case series. Therefore, optimal management of regional lymph nodes for high-risk tumors remains unclear.

Sentinel lymph node biopsy (SNLB) is a common procedure utilized in multiple oncologic surgeries, especially dermatology. SLNB is recommended for aggressive skin cancers including melanoma and Merkel cell carcinoma. There is limited data on the utility of SLNB in nonmelanoma skin cancers, including cutaneous SCC. To date, there have been no prospective trials and current data comes from small retrospective studies. Therefore, the impact of SLNB on management and outcomes with high-risk cSCC remains unknown. Therefore, the impact of SLNB on cSCC remains unclear. The purpose of this study is to evaluate the rate of occult metastasis utilizing sentinel lymph node biopsy in clinically node-negative intermediate and high-risk cSCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old at the time of informed consent
* Ability to provide written informed consent and HIPAA authorization
* Primary or recurrent invasive cutaneous squamous cell carcinoma of the head or neck, clinically staged T2-T4 based on AJCC staging
* Clinically and radiographically regional node-negative (no evidence of regional lymph node metastasis or distant metastasis)
* Able to undergo general anesthesia for sentinel lymph node biopsy
* Able to undergo CT scan with contrast or MRI with contrast
* Undergo surgical resection (Moh's or micrographic resection or standard excision with sentinel lymph node biopsy) within 8 weeks of imaging

Exclusion Criteria:

* Clinical evidence of satellite lesions, in-transit, regional nodal or distant metastases
* Known biopsy proven synchronous primary cutaneous squamous cell carcinoma
* Pregnant patients
* Patients unable to undergo general anesthesia
* Patient unable to receive contrasted imaging studies
* Patient unable to receive and/or allergic to 99m-Technetium sulfur colloid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of metastasis | Baseline
  Incidence of occult metastasis in cT2-4N0 cutaneous squamous cell carcinoma (cSCC) of the head and neck by measuring the number of patients with positive sentinel lymph node biopsies.

SECONDARY OUTCOMES:
Evaluate the tumor variables | Baseline to 1 year
  Evaluate the tumor variables associated with occult metastasis using Fisher's exact tests for characteristics with categorical data and using logistic regression for characteristics with continuous data. (Tumor characteristics will be evaluated for their association with metastasis. Analyses will evaluate each of the characteristics individually using Fisher's exact tests for characteristics with categorical data and using logistic regression for characteristics with continuous data. No multivariable models will be assessed due to the small number of expected patients with metastasis. A 5% significance level will be used for all tests.)
Evaluate the gene profile via validated 40-gene expression profile (40-GEP) to identify common mutations associated with high-risk tumors characteristics. | Baseline up to 1 year after reoccurrence occurs
  Regional recurrence and distant metastasis confirmed by clinical, pathologic and radiographic evidence of metastasis.
Evaluate the gene profile of tumor | Baseline to 1 year
  Evaluate the gene profile via validated 40-gene expression profile (40-GEP) to identify common mutations associated with high-risk tumors characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Yesensky, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No